CLINICAL TRIAL: NCT06184373
Title: Early Investigation of Glucose Monitoring After Gestational Diabetes (ENGAGED): Utility and Acceptability of Continuous Glucose Monitoring in the Early Postpartum Period After Gestational Diabetes Mellitus
Brief Title: Early Investigation of Glucose Monitoring After Gestational Diabetes Pilot
Acronym: ENGAGED
Status: Recruiting | Type: Observational
Sponsor: Ohio State University (Other)
Collaborators: DexCom, Inc. (Industry)
Responsible Party: Principal Investigator, Rachel D'Amico, Assistant Professor, Ohio State University
Other Study IDs: 2023H0066
Record Dates: First submitted 2023-12-14; First posted 2023-12-28 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Gestational Diabetes; Hyperglycemia
MeSH Terms: conditions — Diabetes, Gestational; Hyperglycemia | interventions — Glucose Tolerance Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Participants: Participants will be recruited at 6-8 weeks postpartum; at that appointment, CGMs will be placed. After wearing the CGM, participants will fill out surveys regarding their experience. At 10-12 weeks postpartum, they will complete the standard of care OGTT as well as complete an interview regarding their experience. At 12 months postpartum, they will complete a blood test to check their hemoglobin A1c.
  Interventions: Device: Continuous glucose monitor; Diagnostic Test: Oral Glucose Tolerance Test; Diagnostic Test: Hemoglobin A1c

INTERVENTIONS:
Device: Continuous glucose monitor — CGMs will be worn for a maximum of 10 days at 6-8 weeks postpartum.
  Other Names: CGM
Diagnostic Test: Oral Glucose Tolerance Test — At 10-12 weeks postpartum, participants will complete an oral glucose tolerance test, which involves drinking a glucose substance and having glucose levels measured a maximum of 3 times.
Diagnostic Test: Hemoglobin A1c — At 11-14 months postpartum, participants will be asked to have their blood drawn to check their hemoglobin A1c to look for signs of developed insulin resistance

SUMMARY:
One third of women with gestational diabetes (GDM), diabetes diagnosed during pregnancy, have abnormal glucose levels within 3 years after pregnancy, but follow up is low. Continuous glucose monitors (CGM), a small sensor inserted under the skin, may be able to screen women with GDM for diabetes risk. The investigators will ask postpartum women to use CGM at 6-8 weeks postpartum and answer surveys about quality of life after wearing the CGM. The investigators will collect data on blood glucose trends for future studies if participants find CGM use acceptable. The investigators hope to learn if CGM could improve postpartum follow up experiences for people with recent GDM.

DETAILED DESCRIPTION:
Gestational diabetes (GDM) is associated with a significantly increased risk of type 2 diabetes, with 1/3 of individuals with GDM developing glucose intolerance in the first 3 years postpartum. The American Diabetes Association recommends a follow up oral glucose tolerance test (OGTT) 4-12 weeks after delivery for all patients with GDM, but rates of follow up screening are as low as 19%. OGTT presents many challenges to postpartum patients, including lengthy visits and the need to fast for at least 8 hours, that likely impact these follow up rates. There is also evidence that many individuals with normal OGTT develop dysglycemia within the first year postpartum, leading to concerns about the diagnostic yield of OGTT. Continuous glucose monitors (CGM) have revolutionized the care of type 1 and 2 diabetes, but its utility in GDM is poorly studied. There are many potential benefits of CGM as a possible GDM postpartum screening, including the ability to transmit data remotely and increased glycemic data, but the impact CGMs have on quality of life postpartum and if they would be acceptable screening methods for patients after delivery has yet to be studied. Our research aims to understand the acceptability and feasibility of CGM for detection of ongoing dysglycemia in the postpartum period in GDM. A sample of 20 postpartum individuals with a history of GDM will have CGMs placed at 6-8 weeks postpartum . Participants will have surveys after the CGM period about CGM impact on quality of life as well as complete a validated glucose monitoring satisfaction survey. They will then complete the standard of care OGTT at 10-12 weeks postpartum and be asked to compare their experience with CGM versus OGTT and which screening method they found preferable. Wear times and study dropout rates will be analyzed for intervention fidelity as a marker of feasibility. The investigators will begin to characterize postpartum glycemia by mean serum glucose, time in range (TIR) and coefficient of variation (CV) as measured by CGM. Glycemic data will be compared to a 12-week OGTT to determine relative sensitivity. This study could determine if CGM may provide a novel screening method for postpartum GDM that is acceptable to patients.

ELIGIBILITY:
Inclusion Criteria:

* Women with a viable singleton intrauterine pregnancy
* Able to understand the study, and having understood, provide written informed consent in English
* Recent pregnancy affected by gestational diabetes

Exclusion Criteria:

* Pregestational Diabetes (Type I or Type II)
* Continued use of diabetes medications (including metformin and insulin) immediately after delivery
* Preterm delivery (< 37 weeks gestation)
* Twin or higher order gestation
* No access to a smartphone
* Unable or unwilling to wear CGM or return for follow up at postpartum mother-infant dyad clinic
* Participation in this trial in a prior pregnancy
* History of skin allergy to adhesive products or CGM

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: We anticipate enrolling a total of 20 participants with a recent pregnancy affected by GDM
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-06-06 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Acceptability of CGM | 15 weeks from enrollment
  As determined by survey
Comparative experience of OGTT and CGM | 15 weeks from enrollment
  As determined by survey

SECONDARY OUTCOMES:
Prevalence and characteristics of dysglycemia in GDM postpartum | 15 weeks from enrollment
  As determined by survey
Lifestyle changes survey | 15 weeks from enrollment
  Breastfeeding practices, changes in diet and physical activity
Medical care | 15 weeks from enrollment
  Number of doctor's visits (both for participant and their infant), prescribed medications

OTHER OUTCOMES:
Infant outcomes | birth outcomes only
  in-hospital medical record review

CONTACTS AND LOCATIONS:
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided